CLINICAL TRIAL: NCT01966952
Title: Centre of Excellence for Treatment of Resistant Hypertension: Establishment and Critical Evaluation of Efficacy, Mechanisms and Safety of Renal Sympathetic Radioablation.
Brief Title: Evaluation of Safety Mechanisms of Renal Radioablation(RSRA)for Uncontrolled Hypertension
Acronym: RSRA
Status: Terminated | Type: Observational
Why Stopped: Simplicity HTN 3 trial did meet safety endpoint, but did not meet efficacy endpoint and withdrew support for their catheter in 2014.
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20130444-01H
Record Dates: First submitted 2013-10-16; First posted 2013-10-22 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Uncontrolled Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Resistant Hypertension: Resistant hypertension as described as; patients with uncontrolled hypertension on 3 or more antihypertensive medications with no secondary causes for hypertension (i.e. hyperaldosteronism, renal artery stenosis)

SUMMARY:
Renal sympathetic radioablation disrupts the nerves by high radiofrequency signal which creates localized heat, eliminates the signal and decrease blood pressure.

The main purpose of this study is to evaluate blood pressure 12 months after radioablation, and to evaluate the short and long-term effects of the renal radioablation on the extent of changes in urine catecholamines level, vascular stiffness, and sympathetic nerve activity as linked with the changes in blood pressure. The study will also evaluate the effect radioablation has on the renal arteries as well as develop teaching sessions for family physicians and other specialists to educate them on this new treatment.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy, safety and selected mechanisms of renal sympathetic radioablation. The primary outcome of this study is change in BP 12 months post treatment as assessed from daytime average of systolic BP from 24-hr ABPM.

In this innovation program, we propose to evaluate the following aspects of renal sympathetic radioablation RSRA in Patients with Resistant HTN:

1. Efficacy:

   Assessment of BP lowering effect in patients with true resistant HTN. In contrast to studies done so far, we will evaluate the true BP lowering effect of RSRA by performance of 24-hr ABPM prior to and at defined time points post procedure. We will screen out pseudohypertension using direct observed therapy. We will employ a rigorous protocol to include only patients with truly resistant HTN. Namely, we will screen for major forms of secondary HTN such as renal artery stenosis, pheochromocytoma, primary hyperaldosteronism, and Cushing's syndrome and exclude these patients from radioablation. We will also address the issue of white coat phenomena as a cause of false diagnosis of resistant HTN by 24-hr ABPM. This innovative approach will ensure a proper evaluation of the BP lowering potential of this method, as patients with secondary forms of HTN may not respond to RSRA. In contrast, those with white coat effect may show gradual improvement in BP control over time unrelated to RSRA.
2. Safety: Imaging of the renal arteries. Our patients will undergo CT angiogram imaging of their renal arteries prior to procedure and at defined time points afterwards. In studies reported so far, imaging of the renal arteries was not standardized. In animals (swines) subjected to RSRA using the same catheter, renal arteries showed fibrosis of 10-25% of the total media and underlying adventitia, with mild disruption of the external elastic lamina. Furthermore, a case report has been published documenting renal artery stenosis within 3 months post RSRA.
3. Education on diagnosis and treatment of resistant HTN. As resistant HTN is frequently misdiagnosed and consequently poorly treated, we will develop teaching sessions for family physicians, general internists, and subspecialists from this LHIN region to make them aware of issues related to diagnosis of true resistant HTN and to educate them on this new option of treatment.
4. Mechanism:

Effects of RSRA on Central Sympathetic Outflow, PWV, and aldosterone will be assessed pre and post RSRA and correlated to (changes in) BP prior to and at defined time points post RSRA.

Clinical relevance:

This is a new method for treatment of patients with resistant HTN. As our team has successfully treated two patients with resistant HTN in June 2012 (as the second team and centre in Canada), TOH/UOHI with experts in Clinical HTN, Nephrology, Interventional Cardiology and Interventional Radiology are uniquely positioned to establish and critically evaluate the suitability of this method for patients from our LHIN region. Pilot data on Pulse Wave Velocity, MSNA and aldosterone by RSRA will shed light on mechanisms involved in BP lowering by RSRA and will be used for the development of grant applications to Canadian peer review funding agencies.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* resistant HTN defined as daytime BP readings above 140/90 mmHg (as assessed from 24-hr ABPM))
* on 4 or more BP lowering drugs

Exclusion Criteria:

* pregnant patients
* Secondary forms of hypertension
* patients with following conditions: eGFR <45 ml/min/1.75 m2,
* active infection,
* known coagulopathies,
* acute coronary syndrome and/or within 6 months post acute coronary event,
* clinically significant arrhythmias,
* within 6 months post stroke/TIA, severe liver disease;
* psychiatric disorders and/or otherwise unable to sign consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be recruited from the Hypetension Units at The Ottawa Hospital and the University of Ottawa Heart Institute. Only patients with uncontrolled hypertension will be eligable.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Blood pressure change post RSRA treatment | 12 months
  Blood pressure(BP)will be assessed post Renal Radiosympathetic radioablation RSRA)by 24-hr Ambulatory blood pressure monitor (ABPM) using the daytime average of systolic BP

SECONDARY OUTCOMES:
efficacy | 1-3-6-&12 months
  changes in daytime average systolic BP by 24-hr ABPM at 1,3, 6,& 12 months post RSRA
  - changes in urinary catecholamines, aldosterone, Pulse wave velocity(PWV), and Muscle Sympathetic Nerve activity (MSNA) at defined time points post treatment.
Safety | 12 months
  Secondary safety outcomes will also include frequency of complications including development of renal artery stenosis post procedure, determined by CT angiogram.

OTHER OUTCOMES:
Education | 24months
  Finally, formal evaluation of our teaching lectures on Diagnosis and Management of Resistant HTN will be part of outlined CMEs.

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Ruzicka, MD, Principal Investigator — The Ottawa Hospital Research Institute
Locations (1):
- The Hypetension Unit of The Ottawa Hospital, Ottawa, Ontario, Canada